CLINICAL TRIAL: NCT02455583
Title: An Assessment of an HIV Prevention Intervention (Project AIM) on Youth Sexual Intentions, Sexual Behaviors and HSV-2 Incidence and Prevalence in Junior Secondary Schools in Eastern Botswana.
Brief Title: An Assessment of an HIV Prevention Intervention (Project AIM) Among Junior Secondary School Students in Eastern Botswana
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Education and Skills Development, Botswana (Unknown); Education Development Center, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6451
Record Dates: First submitted 2015-01-06; First posted 2015-05-28 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: HIV prevention; Sexual activity biomarker; Youth; Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): All Form 1 learners at 25 of the 50 schools will receive HIV prevention sessions from the Botswana life skills education program for junior secondary school students called LIVING.
- Intervention (Experimental): Form 1 learners at the 25 intervention schools will receive the Project AIM intervention and LIVING (standard of care).
  Interventions: Behavioral: Project AIM (Adult Identity Mentoring)

INTERVENTIONS:
Behavioral: Project AIM (Adult Identity Mentoring) — Project AIM consists of 14 sessions that are delivered twice a week. Each session is 40 minutes long.
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine the effectiveness of an HIV prevention intervention called Project AIM (Adult Identity Mentoring) to delay onset of sexual activity and reduce sexual risk behaviors among students (approximate ages 12- 17 years) in junior secondary schools (Form 1 - 3) in Eastern Botswana.

DETAILED DESCRIPTION:
Few behavioral intervention models exist that focus on pre-sexually active adolescents in high-prevalence environments. As a result, there is a paucity of scientific research on HIV education models that impact risk factors among pre-sexual adolescents or that address the underlying causes and contextual factors associated with the sexual risk behaviors that leave adolescents vulnerable to HIV infection. Project AIM (Adult Identity Mentoring) is an evidence-based youth development HIV prevention intervention designed for youth ages 11-14 years. The goals of Project AIM are to provide youth with the motivation to enact safe choices and to address social barriers to sexual risk prevention such as hopelessness, peer pressure, and risk opportunities in low income environments. Results of a United States (U.S.)-based behavioral study have demonstrated a positive effect in reducing sexual intentions and increasing sexual abstinence. Project AIM has not previously been evaluated for use in an African context.

The purpose of this 50 site, stratified, cluster, randomized control trial is to examine the efficacy of Project AIM to delay onset of sexual activity and reduce sexual risk behaviors among students (approximate ages 12- 17 years) in junior secondary schools (JSS) in Eastern Botswana.The study will involve enrolling a longitudinal cohort consisting of Form 1 students who will be randomized to either the intervention (Project AIM) or control condition and followed from the start of the Form 1 year to the end of the Form 3 year.

Outcomes will be assessed through participant self-report of sexual risk behavior and HSV-2 testing as a biomarker of self-reported sexual activity. Participants will complete a behavioral survey three times (baseline, 12 months, and 24 months) and HSV-2 testing two times (baseline and 24 months).

Effective implementation of Project AIM as part of the school health curriculum in Botswana would provide an evidence-based, in-school program option to aid and inform HIV prevention efforts for young adolescents across southern Africa. Implementation of the program will also build on existing programmatic efforts and infrastructure and attempt to demonstrate how the addition of an evidence-based, multi-component HIV prevention program will strengthen current youth HIV prevention policies and programming. In addition, rates of herpes simplex virus type 2 (HSV-2) from the study will provide the region with sexual risk behavior data and HSV-2 prevalence estimates for young adolescents in Eastern Botswana, which can inform public health recommendations as well as national policies for sexual/reproductive health and education among this population.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in Form 1 at one of the 50 selected schools (longitudinal cohort)
* Fluent and literate in English or Setswana
* Able and willing to provide written informed assent (age 17 or under) or informed consent (age 18 and over)
* Parent/guardian provides permission (if age 17 or under) for child to participate

Exclusion Criteria:

- All youth who meet the inclusion criteria may fully participate in the study. No sub-segments of the population will be excluded from participation. Individual students may be excluded from participation by school or study staff due to circumstances in which participation is deemed to not be in the best interest of the student, such as excessive emotional distress.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4732 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Difference in HSV-2 incidence between the intervention and control arm | Baseline and 24 months

SECONDARY OUTCOMES:
Self-reported sexual and sexual risk-related behavior measured by sexual initiation, number of sexual partners and frequency of alcohol use, sexual intercourse, and condom use | Longitudinal Cohort: baseline, 12 months, and 24 months
Sexual thoughts measured by frequency of thoughts about engaging in sexual activity | Longitudinal Cohort: baseline, 12 months, and 24 months
Attitudes towards education and frequency of thoughts and feelings about the future and hopelessness | Longitudinal Cohort: baseline, 12 months, and 24 months
Attitudes towards partner concurrency, transactional sex, and sexual risk communication with a partner | Longitudinal Cohort: baseline, 12 months, and 24 months
Intention to engage in sexual activity | Longitudinal Cohort:baseline, 12 months, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim S Miller, PhD, Principal Investigator — Centers for Disease Control and Prevention; Nontobeko S Tau, Principal Investigator — Botswana: Minsitry of Education and Skills Development
Locations (1):
- 50 Junior Secondary schools, Multiple Locations, Eastern Botswana, Botswana

REFERENCES:
- [Background] Clark LF, Miller KS, Nagy SS, Avery J, Roth DL, Liddon N, Mukherjee S. Adult identity mentoring: reducing sexual risk for African-American seventh grade students. J Adolesc Health. 2005 Oct;37(4):337. doi: 10.1016/j.jadohealth.2004.09.024. PMID 16182145